CLINICAL TRIAL: NCT02895347
Title: Proficiency Based Robotics Training Curriculum: Skill Acquisition & Transferability of Skills
Brief Title: Proficiency Based Robotics Training Curriculum: Skill Acquisition & Transferability of Skills to Live Porcine Models
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 111547
Record Dates: First submitted 2016-09-06; First posted 2016-09-09 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2016-09

CONDITIONS: Medical Students Naive to Surgical Robotics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Participants in the Control Group (CG) were asked to attend an orientation reviewing the study. Three weeks later they returned and were filmed timed completing a suturing activity on the porcine model.
- Experimental Group (Experimental): Participants in the Experimental Group (EG) were asked to attend an orientation reviewing the study. Then they were instructed to complete 4 activities on the dvSS ® that modeled suturing techniques in minimally invasive robotics-assisted surgery. EG participants repeated these 4 activities over a period of 2 weeks until they reached proficiency (91%) in all 4 activities. 4. Participants were asked to return where they were filmed and timed completing a suturing activity on the porcine model.
  Interventions: Behavioral: Surgical Simulation Practice Modules

INTERVENTIONS:
Behavioral: Surgical Simulation Practice Modules — The surgical simulation practice modules simulate surgical settings for suturing.
  Arms: Experimental Group

SUMMARY:
The goal of the project is to define the optimal learning environment and protocol for dvSS® simulation activities using medical students as robotic-naïve research participants.

DETAILED DESCRIPTION:
The goal of the project is to define the optimal learning environment and protocol for dvSS® simulation activities using medical students as robotic-naïve research participants. The investigators propose to accomplish this goal through the following aims:

Specific Aim #1: to investigate the total training time and the total number of repetitions required for participants to achieve proficiency (as defined on the dvSS® as 91%) for each of the selected exercises in selected dVSS activities.

Specific Aim #2: to measure the transferability of skills acquired through a robotic simulation to live porcine models compared to nonintervention controls. The study will compare the effect of training with the dVSS to similar nonintervention controls by grading a suturing procedure on a live porcine model.

Findings generated from this study will provide new insight into the efficacy of the dVSS as a simulation- based training tool for medical practitioners. Collectively, this work will build upon the narrow knowledge base on how to develop a nationally accredited simulation-based robotics curriculum.

This study undoubtedly furthers the GWU SMHS mission of education, research, and healing. The study seeks to understand the learning curve students can achieve by simulation-based training and then to directly apply that training to a safe in vivo model in order to determine training interventions that can inform a robotic curriculum both locally at GWU and throughout the country. Additionally, this study is innovative in that it is the first of its kind to correlate skills acquired on a robotic-simulation gynecology based tool to a live porcine model. It seeks to enhance the current GWU GYN robotics- curriculum and assist with the development of a specific curriculum within the next year. Although the immediate goal is for planning toward a gynecology robotic curriculum, results of this study could also inform development of robotic programs in other disciplines such as general surgery and urology. Considering, the limited development of simulation-based robotics curriculum, further refining the curriculum would allow GWU to continue "to be globally recognized as a medical center that embraces the challenge of…transforming health care, and expanding research to enrich and improve the lives of those [served]." It also serves to "leverage the SMHS brand to enhance opportunities for recognition, distinction..& marketing." Preparing a generation of well-trained and confident gynecologic surgeons will allow providers to administer safe care to women.

ELIGIBILITY:
Inclusion Criteria:

* medical & physician assistant students at George Washington University with no prior experience using a surgical robot

Exclusion Criteria:

* medical & physician assistant students at George Washington University with prior experience using a surgical robot
* students not enrolled in the medical or physician assistant program at George Washington University

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-12; Primary Completion 2016-03 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- George Washington University Medical Faculty Associates, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
Results will be submitted for Association of Processors of Gynecology and Obstetrics Annual Meeting as well as to journals for publication.

REFERENCES:
- [Background] Advincula AP, Wang K. Evolving role and current state of robotics in minimally invasive gynecologic surgery. J Minim Invasive Gynecol. 2009 May-Jun;16(3):291-301. doi: 10.1016/j.jmig.2009.03.003. PMID 19423061
- [Background] Sheth SS, Fader AN, Tergas AI, Kushnir CL, Green IC. Virtual reality robotic surgical simulation: an analysis of gynecology trainees. J Surg Educ. 2014 Jan-Feb;71(1):125-32. doi: 10.1016/j.jsurg.2013.06.009. Epub 2013 Jul 12. PMID 24411435
- [Background] Gobern JM, Novak CM, Lockrow EG. Survey of robotic surgery training in obstetrics and gynecology residency. J Minim Invasive Gynecol. 2011 Nov-Dec;18(6):755-60. doi: 10.1016/j.jmig.2011.08.004. PMID 22024262
- [Background] Brenot K, Goyert GL. Impact of robotic surgery on obstetric-gynecologic resident training. J Reprod Med. 2009 Nov-Dec;54(11-12):675-7. PMID 20120900
- [Background] Hung AJ, Zehnder P, Patil MB, Cai J, Ng CK, Aron M, Gill IS, Desai MM. Face, content and construct validity of a novel robotic surgery simulator. J Urol. 2011 Sep;186(3):1019-24. doi: 10.1016/j.juro.2011.04.064. Epub 2011 Jul 23. PMID 21784469
- [Background] Kenney PA, Wszolek MF, Gould JJ, Libertino JA, Moinzadeh A. Face, content, and construct validity of dV-trainer, a novel virtual reality simulator for robotic surgery. Urology. 2009 Jun;73(6):1288-92. doi: 10.1016/j.urology.2008.12.044. Epub 2009 Apr 10. PMID 19362352
- [Background] Stegemann AP, Ahmed K, Syed JR, Rehman S, Ghani K, Autorino R, Sharif M, Rao A, Shi Y, Wilding GE, Hassett JM, Chowriappa A, Kesavadas T, Peabody JO, Menon M, Kaouk J, Guru KA. Fundamental skills of robotic surgery: a multi-institutional randomized controlled trial for validation of a simulation-based curriculum. Urology. 2013 Apr;81(4):767-74. doi: 10.1016/j.urology.2012.12.033. Epub 2013 Feb 26. PMID 23484743
- [Background] Stefanidis D, Wang F, Korndorffer JR Jr, Dunne JB, Scott DJ. Robotic assistance improves intracorporeal suturing performance and safety in the operating room while decreasing operator workload. Surg Endosc. 2010 Feb;24(2):377-82. doi: 10.1007/s00464-009-0578-0. Epub 2009 Jun 18. PMID 19536599
- [Background] Aghazadeh MA, Jayaratna IS, Hung AJ, Pan MM, Desai MM, Gill IS, Goh AC. External validation of Global Evaluative Assessment of Robotic Skills (GEARS). Surg Endosc. 2015 Nov;29(11):3261-6. doi: 10.1007/s00464-015-4070-8. Epub 2015 Jan 22. PMID 25609318

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 40 subjects who consented to participate in the study, 4 subjects failed to complete study procedures and dropped out of the study. Reason for this included inability to attend the final assessment and subjects unwilling to perform the final study assessment on a live porcine model.
Groups:
- Control Group: Participants in the Control Group (CG) were asked to attend an orientation reviewing the study. Three weeks later participants returned and were filmed timed completing a suturing activity on the porcine model.
- Experimental Group: Participants in the Experimental Group (EG) were asked to attend an orientation reviewing the study. Then participants were instructed to complete 4 activities on the dvSS ® that modeled suturing techniques in minimally invasive robotics-assisted surgery. EG participants repeated these 4 activities over a period of 2 weeks until proficiency (91%) in all 4 activities was reached. Participants were asked to return and were filmed and timed completing a suturing activity on the porcine model.
Period: Overall Study
Arm/Group | Control Group | Experimental Group
Started | 20 | 20
Completed | 17 | 19
Not Completed | 3 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Experimental Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Full Range); unit: years] | 25 [22 to 40] | 25 [22 to 40] | 25 [22 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 13 | 9 | 22
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Global Evaluative Assessment of Robotic Skills (GEARS) Scale
Description: GEARS is a validated assessment tool for grading overall technical proficiency for robotic surgery. The overall proficiency score is a composite score of five different measures: depth perception, bimanual dexterity, efficiency, force sensitivity, and robotic control. Each of these subscale scores are graded 1-5, with 1 being poor and 5 being excellent. The total score is the summation of the scores from each of the five subscales and ranges from 5 to 25.
Time Frame: Three weeks after orientation
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 17 | 19
units on a scale | 15.25 (3.38) | 15.37 (2.51)

2. Primary Outcome: Amount Time to Suture
Description: time, measured in minutes, it took each participant to perform the suturing activity
Time Frame: Three weeks after orientation
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 17 | 19
minutes | 9.9 (2.07) | 9.2 (2.65)

3. Primary Outcome: Amount of Time to Achieve Proficiency
Description: time, measured in minutes, it took each participant in the intervention group to achieve surgical proficiency on the robotic simulator.
Time Frame: assessed after the orientation and prior to the three week date for the final suturing assessment
Measure: Mean (Full Range); unit: minutes
Arm/Group | Experimental Group
Number analyzed (Participants) | 19
minutes | 116 [53 to 209]

ADVERSE EVENTS:
Time Frame: subjects were monitored for adverse events (AEs) throughout the entire duration of study participation (a total of 3 weeks)
Arm/Group | Control Group | Experimental Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No